CLINICAL TRIAL: NCT01853228
Title: Phase 1-2 Safety and Efficacy Study of DACOGEN in Sequential Administration With Cytarabine in Children With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: A Study of Decitabine (DACOGEN) in Sequential Administration With Cytarabine in Children With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: EMA/PDCO acknowledged that available results from this study do not support further clinical studies in relapsed/refractory AML paediatric patients.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR102071; DACOGENAML2004 (Other: Janssen Research & Development, LLC); 2013-000390-70 (EudraCT Number)
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Relapsed or refractory acute myeloid leukemia; Children; Decitabine; DACOGEN; Cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Decitabine and cytarabine (Experimental)
  Interventions: Drug: Phase1 and Phase 2: decitabine; Drug: Phase 1: cytarabine; Drug: Phase 2: cytarabine

INTERVENTIONS:
Drug: Phase1 and Phase 2: decitabine — 20 mg/m2 administered by intravenous infusion over 1 hour once daily for 5 consecutive days (Day 1 to Day 5 of 28-day cycle)
Drug: Phase 1: cytarabine — 1 g/m2, 2 g/m2, and 1.5 g/m2 dose levels administered by intravenous infusion over 4 hours daily for 5 consecutive days (Day 8 to Day 12 of 28-day cycle) for the determination of the maximum tolerated dose
Drug: Phase 2: cytarabine — Phase 1 maximum tolerated dose administered by intravenous infusion over 4 hours daily for 5 consecutive days (Day 8 to Day 12 of 28-day cycle)

SUMMARY:
The purpose of this study is to examine the safety and efficacy of decitabine in sequential administration with cytarabine in children with relapsed or refractory acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known) study to evaluate safety, efficacy, and pharmacokinetics (study of what the body does to a drug) of decitabine in sequential administration with cytarabine in children with relapsed or refractory AML. The study will determine the maximum tolerated dose of cytarabine that can be given following decitabine (Phase 1) and the response rate to this combination (Phase 2). Participants may enter a continuation phase of single agent-decitabine infusions for as long as such treatment would be considered beneficial. Serial pharmacokinetic samples will be collected and safety and efficacy will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of acute myeloid leukemia (AML) according to the World Health Organization (WHO) classification
* Diagnosis of AML which has relapsed or is refractory to standard of care and no curative therapy exists
* Karnofsky or Lansky score of at least 50
* Must be recovered from acute toxicity of any prior treatment
* Must have adequate organ function according to protocol-defined criteria
* Agrees to protocol-defined use of effective contraception
* Female participants of childbearing potential must have a negative serum or urine pregnancy test at Day 1 of Cycle 1

Exclusion Criteria:

* Prior treatment with decitabine or azacitidine
* Acute promyelocytic leukemia (M3 subtype in the French-American-British [FAB] classification system)
* CNS3 disease
* acute myeloid leukemia (AML) associated with congenital syndromes such as Down syndrome, Fanconi anemia, Bloom syndrome, Kostmann syndrome or Diamond-Blackfan anemia, or bone marrow failure associated with inherited syndromes
* White blood cell count greater than 40x10^9 cells/liter(L)
* Known allergies, hypersensitivity, or intolerance to decitabine or cytarabine or their excipients
* Contraindications to the use of cytarabine per local prescribing information or prior adverse reactions to cytarabine which would prevent further use
* Currently enrolled in the treatment phase of an interventional investigational study
* Female who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 3 months after the last dose of study drug (however, the period after which it becomes safe to become pregnant after the last dose of treatment is not known)
* Male who plans to father a child while enrolled in this study or within 3 months after the last dose of study drug
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient or that could prevent, limit, or confound the protocol-specified assessments
* Any social or medical condition that in the investigator's opinion renders the participant unfit for study participation
* History of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease
* History of human immunodeficiency virus (HIV) antibody positive

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (17):
- Ghent, Belgium
- Copenhagen Ø, Denmark
- France (3):
  - Paris
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (4):
  - Essen
  - Hamburg
  - Hanover
  - Stuttgart
- Rotterdam, Netherlands
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia
- United Kingdom (4):
  - Birmingham
  - Cambridge
  - Glasgow
  - Sutton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 17 participants were enrolled in the study. 16 participants were enrolled in Phase 1 (9 participants in Cohort 1 and 7 participants in Cohort 2). 7 participants of Cohort 2 continued to Phase 2. One additional participant was enrolled in Phase 2 of the study, making a total of 8 participants evaluable in Phase 2.
Groups:
- Cohort 1: Decitabine 20 mg/m^2 + Cytarabine 1 g/m^2: Participants received decitabine 20 milligram per square meter (mg/m^2) by intravenous infusion over 1 hour once daily for 5 consecutive days (Day 1 to Day 5 of each 28-day cycle). In addition, participants received cytarabine 1 gram per square meter (g/m^2) dose levels administered by intravenous infusion over 4 hours daily for 5 consecutive days (Day 8 to Day 12 of each 28-day cycle) for the determination of the maximum tolerated dose in Cohort 1 of Phase 1.
- Cohort 2: Decitabine 20 mg/m^2 + Cytarabine 2 g/m^2: Participants received decitabine 20 mg/m^2 by intravenous infusion over 1 hour once daily for 5 consecutive days (Day 1 to Day 5 of each 28-day cycle) in Phase 1 and Phase 2. In addition, participants received cytarabine 2 g/m^2 dose levels administered by intravenous infusion over 4 hours daily for 5 consecutive days (Day 8 to Day 12 of each 28-day cycle) for the determination of the maximum tolerated dose in Cohort 2 of Phase 1. Participants who completed Phase 1 were continued in Phase 2 and received cytarabine at MTD determined in Phase 1 (2 g/m^2) by intravenous infusion over 4 hours daily for 5 consecutive days (Day 8 to Day 12 of each 28-day cycle).
Period: Phase 1
Arm/Group | Cohort 1: Decitabine 20 mg/m^2 + Cytarabine 1 g/m^2 | Cohort 2: Decitabine 20 mg/m^2 + Cytarabine 2 g/m^2
Started | 9 | 7
Completed | 0 | 7 (Participants who completed Phase 1 moved to Phase 2.)
Not Completed | 9 | 0
Not completed — Lack of Efficacy | 8 | 0
Not completed — Other | 1 | 0
Period: Phase 2
Arm/Group | Cohort 1: Decitabine 20 mg/m^2 + Cytarabine 1 g/m^2 | Cohort 2: Decitabine 20 mg/m^2 + Cytarabine 2 g/m^2
Started | 0 | 8 (1 additional participant was enrolled, making total of 8 participants evaluable in Phase 2.)
Completed | 0 | 0
Not Completed | 0 | 8
Not completed — Physician Decision | 0 | 1
Not completed — Proceed To Transplant | 0 | 3
Not completed — Lack of Efficacy | 0 | 4

BASELINE CHARACTERISTICS:
Population: Population included all enrolled participants in Phase 1 and Phase 2.
Groups:
- Dacogen + Cytarabine: Participants received decitabine 20 milligram per square meter (mg/m^2) by intravenous infusion over 1 hour once daily for 5 consecutive days (Day 1 to Day 5 of each 28-day cycle) in Phase 1 and Phase 2. In addition, participants received cytarabine 1 gram per square meter (g/m^2) (Cohort 1) and 2 g/m^2 (Cohort 2) dose levels administered by intravenous infusion over 4 hours daily for 5 consecutive days (Day 8 to Day 12 of each 28-day cycle) for the determination of the maximum tolerated dose in Phase 1. The maximum tolerated dose identified in Phase 1 was administered by intravenous infusion over 4 hours daily for 5 consecutive days (Day 8 to Day 12 of a 28-day cycle) in Phase 2.
Arm/Group | Dacogen + Cytarabine
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: months] | 73.3 (46.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 1
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 1
  Denmark | 2
  France | 4
  Germany | 1
  Netherlands | 1
  Spain | 4
  United Kingdom | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) of Cytarabine
Description: The maximum tolerated dose (MTD) for cytarabine was based on the number of participants experiencing a dose-limiting toxicity (DLT) by the end of Cycle 1. A non-hematological DLT was defined as: any Grade >=3 toxicity that persists for greater than (>) 5 days or any Grade 2 toxicity that persists for >7 days and that is intolerable to the participant. A hematological DLT was defined as Grade 4 neutropenia or thrombocytopenia due to a hypoplastic bone marrow at Day 42, in the absence of malignant infiltration. The nominal duration of each cycle was 28 days. However, participants who had not experienced bone marrow recovery at Day 28 were followed up to Day 42. Failure of marrow recovery (improvement to Grade 3) by Day 42 was considered a DLT. The maximum duration of Cycle 1 was therefore 42 days.
Time Frame: Cycle 1 (42 days)
Population: Population included participants who experienced a DLT by the end of Cycle 1.
Measure: Number; unit: gram per square meter
Groups:
- Decitabine (Dacogen) + Cytarabine: Participants received decitabine 20 milligram per square meter (mg/m^2) by intravenous infusion over 1 hour once daily for 5 consecutive days (Day 1 to Day 5 of each 28-day cycle) in Phase 1 and Phase 2. In addition, participants received cytarabine 1 gram per square meter (g/m^2) and 2 g/m^2 dose levels administered by intravenous infusion over 4 hours daily for 5 consecutive days (Day 8 to Day 12 of each 28-day cycle) for the determination of the maximum tolerated dose in Phase 1. The maximum tolerated dose identified in Phase 1 was administered by intravenous infusion over 4 hours daily for 5 consecutive days (Day 8 to Day 12 of a 28-day cycle) in Phase 2.
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 6
gram per square meter | 2

2. Secondary Outcome: Phase 1 and 2: Maximum Plasma Concentration (Cmax) of Decitabine
Description: Cmax is the maximum observed plasma concentration of Decitabine.
Time Frame: Cycle 1 (28 days) Day 5: pre-infusion, 0.5 hour during infusion, end of infusion and at 5 min, 0.5 hour, 1 hour, and 2 hour after end of infusion
Population: Population included all enrolled participants in this study assessed for PK. Pharmacokinetic analysis was planned to be reported for the overall participants including Phase 1 and 2. Here 'n' signifies number of participants analyzed for specified category.
Measure: Median (Full Range); unit: nanogram per milliliter (ng/mL)
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 17
nanogram per milliliter (ng/mL)
  > 1 month to <= 2 years: number analyzed (Participants) | 1
  > 1 month to <= 2 years | 118.4 [17.6 to 1621]
  > 2 to <= 6 years: number analyzed (Participants) | 9
  > 2 to <= 6 years | 123.1 [15.6 to 1012]
  > 6 to <= 12 years: number analyzed (Participants) | 5
  > 6 to <= 12 years | 148.7 [16.5 to 1415]
  > 12 to <= 16 years: number analyzed (Participants) | 2
  > 12 to <= 16 years | 151.4 [19.1 to 1303]

3. Primary Outcome: Phase 1 and 2: Total Clearance of Decitabine
Description: Total clearance of drug after intravenously administration was calculated as: dose/area under the plasma concentration-time curve.
Time Frame: Cycle 1 (28 days) Day 5: pre-infusion, 0.5 hour during infusion, end of infusion and at 5 minute (min), 0.5 hour, 1 hour, and 2 hour after end of infusion
Population: Population included all enrolled participants in this study assessed for pharmacokinetics (PK). Pharmacokinetic analysis was planned to be reported for the overall participants including Phase 1 and 2. Here 'n' signifies number of participants analyzed for specified category.
Measure: Median (Full Range); unit: liter per hour per square meter
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 17
liter per hour per square meter
  >1 month to less than or equal to (<=) 2 years: number analyzed (Participants) | 1
  >1 month to less than or equal to (<=) 2 years | 160.6 [11.7 to 942.3]
  Greater than (>) 2 to <= 6 years: number analyzed (Participants) | 9
  Greater than (>) 2 to <= 6 years | 152.1 [19.5 to 1061]
  > 6 to <= 12 years: number analyzed (Participants) | 5
  > 6 to <= 12 years | 125.9 [13.3 to 951.3]
  > 12 to <= 16 years: number analyzed (Participants) | 2
  > 12 to <= 16 years | 123.2 [11.4 to 832.6]

4. Secondary Outcome: Phase 1 and 2: Area Under the Plasma Concentration-Time Curve (AUC) of Decitabine
Description: AUC is the area under the plasma concentration-time curve of decitabine.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 17
nanogram*hour per milliliter (ng*h/mL)
  > 1 month to <= 2 years: number analyzed (Participants) | 1
  > 1 month to <= 2 years | 124.8 [21.3 to 1708]
  > 2 to <= 6 years: number analyzed (Participants) | 9
  > 2 to <= 6 years | 131.5 [19.3 to 1028]
  > 6 to <= 12 years: number analyzed (Participants) | 5
  > 6 to <= 12 years | 158.9 [21.0 to 1508]
  > 12 to <= 16 years: number analyzed (Participants) | 2
  > 12 to <= 16 years | 162.4 [24.2 to 1747]

5. Secondary Outcome: Phase 2: Duration of Response
Description: Duration of response is defined as weeks from date of first response to date of first relapse or date of death.
Time Frame: From time of response to relapse, study completion/withdrawal, or death, whichever comes first, for up to approximately 3 years 10 months
Population: Population included all enrolled participants who achieved CR or CRi response in Phase 2. There was insufficient data to perform Kaplan Meier analysis, therefore individual data for each evaluable participant was reported.
Measure: Number; unit: weeks
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 2
weeks
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 44.6
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 6.3

6. Secondary Outcome: Phase 2: Overall Response Rate
Description: Overall response rate is defined as percentage of participants with complete remission (CR) +complete remission with incomplete blood count recovery (CRi)+partial remission (PR) per IWG Criteria. CRi: morphologic CR with residual neutropenia (less than [<] 1,000/microliter) or thrombocytopenia <100,000/microliter). CR is defined as morphologic leukemia-free state, with less than 5 percentage (%) blasts in aspirate sample with marrow spicules and with a count of greater than or equal to (>=) 200 nucleated cells, plus absolute neutrophil count (ANC) greater than (>) 1,000/ microliter platelet count of >100,000/microliter and participant must be independent of transfusions for a minimum of 1 week before each marrow assessment. PR: all the same hematologic values of a CR, but with a decrease of >=50% of the percentage of blasts to 5% to 25% in the bone marrow aspirate.
Time Frame: Up to approximately 3 years 10 months
Population: Population included all enrolled participants evaluable in Phase 2.
Measure: Number; unit: Percentage of participants
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 8
Percentage of participants | 37.5

7. Secondary Outcome: Phase 1 and 2: Overall Survival (OS)
Description: OS is defined as the time from the date of first dose of study drug to date of death from any cause. If the participant is alive or the vital status is unknown, the participant will be censored at the date the participant will be last known to be alive.
Time Frame: From enrollment to death or withdrawal, whichever comes first, for up to approximately 3 years 10 months
Population: Population included all enrolled participants in Phase 1 and Phase 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 17
months | 5.1 [3.1 to 11.4]

8. Secondary Outcome: Phase 1 and 2: Event-Free Survival
Description: Event free survival is defined as the time from first dose of study drug to relapse from CR, death, or second malignancy for participants who achieved CR. CR is defined as morphologic leukemia-free state, with less than 5 percentage (%) blasts in aspirate sample with marrow spicules and with a count of greater than or equal to (>=) 200 nucleated cells, plus absolute neutrophil count (ANC) greater than (>) 1,000/ microliter platelet count of >100,000/microliter and participant must be independent of transfusions for a minimum of 1 week before each marrow assessment.
Time Frame: From enrollment to progression/relapse, death, or withdrawal, whichever comes first, for up to approximately 3 years 10 months
Population: Population included all enrolled participants in Phase 1 and Phase 2.
Measure: Median (Full Range); unit: days
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 17
days | 1 [1 to 348]

9. Secondary Outcome: Phase 1 and 2: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are defined as adverse events with onset or worsening on or after date of first dose of study treatment. An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Approximately 3 years 10 months
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug (DACOGEN). This outcome measure was planned to be reported for the overall participants including Phase 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 17
Participants | 17

10. Primary Outcome: Phase 1 and 2: Volume of Distribution at Steady-State (Vss) of Decitabine
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: liter per square meter
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 17
liter per square meter
  > 1 month to <= 2 years: number analyzed (Participants) | 1
  > 1 month to <= 2 years | 35.9 [2.7 to 558.4]
  > 2 to <= 6 years: number analyzed (Participants) | 9
  > 2 to <= 6 years | 36.5 [1.4 to 535.0]
  > 6 to <= 12 years: number analyzed (Participants) | 5
  > 6 to <= 12 years | 31.8 [2.0 to 645.8]
  > 12 to <= 16 years: number analyzed (Participants) | 2
  > 12 to <= 16 years | 35.9 [2.8 to 578.9]

11. Primary Outcome: Phase 2: Percentage of Participants Who Achieved CR or CRi at Cycle 1 Day 28
Description: Response rate (percentage of participants who achieved CR or CRi) was measured using international working group (IWG) criteria. Response rate is defined as complete remission (CR) or complete remission with incomplete blood count recovery (CRi) in children with relapsed or refractory acute myeloid leukemia. CRi is defined as morphologic CR with residual neutropenia (less than [<] 1,000/microliter) or thrombocytopenia <100,000/ microliter). CR is defined as morphologic leukemia-free state, with less than 5 percentage (%) blasts in aspirate sample with marrow spicules and with a count of greater than or equal to (>=) 200 nucleated cells, plus absolute neutrophil count (ANC) greater than (>) 1,000/ microliter, platelet count of >100,000/microliter and participant must be independent of transfusions for a minimum of 1 week before each marrow assessment.
Time Frame: Cycle 1 (28 days) Day 28
Population: Population included all enrolled participants evaluable in Phase 2. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 5
percentage of participants | 20

12. Primary Outcome: Phase 2: Percentage of Participants Who Achieved CR or CRi at Cycle 2 Day 28
Description: as for outcome 11
Time Frame: Cycle 2 (28 days) Day 28
Population: Population included all enrolled participants evaluable in Phase 2. Here 'N' signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 3
percentage of participants | 66.7

13. Primary Outcome: Phase 2: Percentage of Participants Who Achieved CR or CRi at End of Study Treatment
Description: as for outcome 11
Time Frame: End of study treatment (approximately 3 years)
Population: Population included all enrolled participants evaluable in Phase 2.
Measure: Number; unit: percentage of participants
Arm/Group | Decitabine (Dacogen) + Cytarabine
Number analyzed (Participants) | 8
percentage of participants | 12.5

ADVERSE EVENTS:
Time Frame: Screening up to end of study (approximately 3 years 10 months)
Description: The safety analysis set included all enrolled participants who received at least 1 dose of study drug (DACOGEN). The AE data was planned to be analyzed separately for Phase 1 (Cohort 1) and combined for participants in Phase 1 (Cohort 2) and Phase 2.
Groups:
- Phase 1 (Cohort 1): Dacogen + Cytarabine: Participants received decitabine 20 milligram per square meter (mg/m^2) by intravenous infusion over 1 hour once daily for 5 consecutive days (Day 1 to Day 5 of each 28-day cycle) in Phase 1. In addition, participants received cytarabine 1 gram per square meter (g/m^2) and 2 g/m^2 dose levels administered by intravenous infusion over 4 hours daily for 5 consecutive days (Day 8 to Day 12 of each 28-day cycle) for the determination of the maximum tolerated dose in Phase 1.
- Phase 1 (Cohort 2) and Phase 2: Dacogen + Cytarabine: Participants received decitabine 20 mg/m^2 by intravenous infusion over 1 hour once daily for 5 consecutive days (Day 1 to Day 5 of a 28-day cycle) in Phase 1 and Phase 2. In addition, participants received cytarabine 2 g/m^2 dose levels administered by intravenous infusion over 4 hours daily for 5 consecutive days (Day 8 to Day 12 of a 28-day cycle) for the determination of the maximum tolerated dose in Cohort 2 of Phase 1 and continued to receive (2 g/m^2) in Phase 2.
Arm/Group | Phase 1 (Cohort 1): Dacogen + Cytarabine | Phase 1 (Cohort 2) and Phase 2: Dacogen + Cytarabine
All-Cause Mortality (participants affected / at risk) | 8/9 | 6/8
Serious Adverse Events (participants affected / at risk) | 4/9 | 4/8
Other Adverse Events (participants affected / at risk) | 9/9 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (Cohort 1): Dacogen + Cytarabine (N=9) | Phase 1 (Cohort 2) and Phase 2: Dacogen + Cytarabine (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Keratitis (Eye disorders) | 0 | 1
Complication Associated with Device (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Lung Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (Cohort 1): Dacogen + Cytarabine (N=9) | Phase 1 (Cohort 2) and Phase 2: Dacogen + Cytarabine (N=8)
Anaemia (Blood and lymphatic system disorders) | 6 | 8
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 5
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4
Tachycardia (Cardiac disorders) | 1 | 1
Conjunctivitis Allergic (Eye disorders) | 1 | 0
Dry Eye (Eye disorders) | 0 | 1
Keratitis (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Anal Inflammation (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 0
Lip Haemorrhage (Gastrointestinal disorders) | 0 | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 3
Tongue Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 5
Asthenia (General disorders) | 0 | 1
Catheter Site Haemorrhage (General disorders) | 1 | 0
Face Oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 6
Cholestasis (Hepatobiliary disorders) | 0 | 2
Hepatocellular Injury (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1
Enterobacter Infection (Infections and infestations) | 1 | 0
Fungal Infection (Infections and infestations) | 1 | 0
Hepatic Infection (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 2 | 0
Paronychia (Infections and infestations) | 1 | 0
Pneumonia Klebsiella (Infections and infestations) | 0 | 1
Pseudomonas Infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0
Adenovirus Test Positive (Investigations) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 3 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Blood Albumin Decreased (Investigations) | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness Postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Device Occlusion (Product Issues) | 1 | 0
Depressed Mood (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Vulvovaginal Inflammation (Reproductive system and breast disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis Atrophic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Butterfly Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Lividity (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The Sponsor terminated the study earlier than planned due to lack of efficacy with 8 evaluable participants in Phase 2 with no clinically meaningful anti-leukemic activity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT01853228/Prot_SAP_000.pdf